CLINICAL TRIAL: NCT01862497
Title: Mechanism of Increased Ambulatory Blood Pressure in Patients With Intradialytic Hypertension and Hemodialysis Controls: A Case Control Study and Crossover Trial Comparing Carvedilol and Prazosin Hydrochloride
Brief Title: Mechanisms of Increased Ambulatory Blood Pressure in Patients With Intradialytic Hypertension
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Peter Van Buren, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 052012-029
Record Dates: First submitted 2013-05-18; First posted 2013-05-24 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Intradialytic Hypertension
Keywords: Intradialytic Hypertension; Hemodialysis; Hypertension; Extracellular Volume; Endothelial Cell Dysfunction; Endothelin 1; Carvedilol
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum collection for measurement of endothelin-1, asymetic dimethylarginine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Carvedilol (for Aim 3 only): Eligible case subjects from aims 1-2 will participate in a randomized crossover study where each subject will receive carvedilol and prazosin for 8 weeks each(under randomized treatment sequence) with a 1 week washout period included in between treatments.
  The first arm will include subjects that are assigned to the randomization sequence: Carvedilol x 8 weeks (titrated up to 50 mg po bid), washout x 1 week, Prazosin x 8 weeks (titrated up to 16 mg daily)
  Interventions: Drug: Carvedilol vs. Prazosin
- Prazosin (for Aim 3 only): Eligible case subjects from aims 1-2 will participate in a randomized crossover study where each subject will receive carvedilol and prazosin for 8 weeks each(under randomized treatment sequence) with a 1 week washout period included in between treatments.
  The first arm will include subjects that are assigned to the randomization sequence: Prazosin x 8 weeks, washout x 1 week, Carvedilol x 8 weeks
  Interventions: Drug: Carvedilol vs. Prazosin

INTERVENTIONS:
Drug: Carvedilol vs. Prazosin

SUMMARY:
The purpose of this study is 1) to determine what physiologic factors (extracellular fluid overload or vasoconstriction) contribute more to increased blood pressure levels between dialysis treatments in hemodialysis patients whose blood pressure increases and decreases during hemodialysis and 2) to determine whether carvedilol provides better control of blood pressure between dialysis treatments than prazosin in patients whose blood pressure increases during dialysis.

ELIGIBILITY:
Inclusion Criteria (for Aims 1 and 2):

* age more than 18 years
* Hypertension defined as systolic blood pressure more than 140 mmHg before dialysis or more than 130 mmHg after dialysis
* For case subjects with intradialytic hypertension: systolic blood pressure increase more than 10 mmHg from pre to post dialysis in at least 4 out of 6 screening treatments
* For control subjects: systolic blood pressure decrease more than 10 mmHg from pre to post dialysis in at least 4 out of 6 screening treatments

Inclusion criteria for Aim 3 includes the case subjects described above.

Exclusion Criteria:

For Aims 1 and 2:

* Hemodialysis vintage less than 1 month
* Amputated arm or leg
* Presence of cardiac defibrillator or pacemaker
* Presence of large metal prosthesis
* Failure to achieve dry weight

For Case subjects participating in Aim 3:

* Patients with a specific indication for beta blocker therapy including systolic heart failure, history of myocardial infarction, history of tachyarrhythmia or angina being managed with beta blocker therapy.
* Patients with contraindications to beta blockade including bradycardia (heart rate less than 60 beats per minute) while not on a pulse lowering drug, severe reactive airway disease, prior intolerance to beta blocker therapy
* Prior intolerance to alpha blocker therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population includes hypertensive hemodialysis patients.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Ratio of Extracellular Body Water to Total Body Water | Expected recruitment is 4-5 years

SECONDARY OUTCOMES:
Change in Endothelin-1 from pre to post dialysis | Expected recruitment is 4-5 years

OTHER OUTCOMES:
Change in Vascular Resistance from pre to post dialysis | Expected recruitment is 4-5 years
Change in Asymmetric Dimethylarginine From pre to post dialysis | Expected recruitment is 4-5 years
Change in Angiotensin II from pre to post dialysis | Expected recruitment is 4-5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Jung J, Jeon-Slaughter H, Nguyen H, Patel J, Sambandam KK, Shastri S, Van Buren PN. Hyperphosphatemia and its relationship with blood pressure, vasoconstriction, and endothelial cell dysfunction in hypertensive hemodialysis patients. BMC Nephrol. 2022 Aug 23;23(1):291. doi: 10.1186/s12882-022-02918-0. PMID 35999520